CLINICAL TRIAL: NCT00023985
Title: Vaccination With Autologous Tumor Lysate-Pulsed Dendritic Cells - Phase I
Brief Title: Vaccine Therapy in Treating Patients With Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Timothy Anderson, MD, Roswell Park Cancer Institute
Purpose: Treatment
Other Study IDs: CDR0000068881; RPCI-RP-9907; NCI-G01-2007
Record Dates: First submitted 2001-09-13; First posted 2003-01-27 (Estimated); Last update posted 2011-03-07 (Estimated); Status verified 2011-03

CONDITIONS: Lung Cancer
Keywords: stage I non-small cell lung cancer; stage II non-small cell lung cancer; stage IIIA non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — FANG vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: autologous tumor cell vaccine
Biological: therapeutic autologous dendritic cells
Procedure: conventional surgery

SUMMARY:
RATIONALE: Vaccines made from a person's tumor cells and white blood cells may make the body build an immune response to kill tumor cells.

PURPOSE: Phase I trial to study the effectiveness of vaccine therapy in treating patients who have non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and feasibility of immunization with autologous tumor lysate-pulsed dendritic cell vaccine in patients with non-small cell lung cancer.
* Determine the immunologic response in patients treated with this vaccine.

OUTLINE: Patients undergo surgery to remove all or most of the gross evidence of tumor. Two months after surgery (or 4 months if chemotherapy and/or radiotherapy are required), patients undergo leukapheresis. Peripheral blood mononuclear cells are isolated and cultured with interleukin-4 and sargramostim (GM-CSF) to generate dendritic cells (DC). DC are then pulsed with tumor lysate prepared from previously removed tumor. Patients receive autologous tumor lysate-pulsed DC vaccine subcutaneously twice, 4 weeks apart.

Patients are followed every 4 months for 2 years, every 6 months for 1 year, and then annually thereafter.

PROJECTED ACCRUAL: A total of 10 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of operable stage IB, II, or IIIA non-small cell lung cancer

  * Tumor diameter of at least 3 cm

PATIENT CHARACTERISTICS:

Age:

* 18 to 75

Performance status:

* ECOG 0-2

Life expectancy:

* At least 3 months

Hematopoietic:

* WBC at least 3,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 2.0 mg/dL
* AST less than 2 times upper limit of normal (ULN)
* Lactate dehydrogenase less than 2 times ULN
* Hepatitis B and C negative

Renal:

* Creatinine no greater than 1.4 mg/dL

Other:

* Positive cell mediated immunity test (i.e., greater than 5 mm induration in 48 hours with purified protein derivative (of tuberculin), candida, and mumps intradermal injection skin test)
* HIV negative
* No active systemic infection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior biological materials

Chemotherapy:

* At least 4 weeks since prior cytotoxic or chemotherapeutic agents
* Concurrent chemotherapy allowed after surgery and before vaccination

Endocrine therapy:

* No concurrent steroid therapy

Radiotherapy:

* At least 4 weeks since prior radiotherapy
* Concurrent radiotherapy allowed after surgery and before vaccination

Surgery:

* See Disease Characteristics

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-01; Primary Completion 2003-07 (Actual); Study Completion 2003-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy M. Anderson, MD, Study Chair — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States